CLINICAL TRIAL: NCT07322107
Title: Observation of Prefrontal Cortex Activation and Electrocardiographic Characteristics in Stroke Patients and Healthy Adults
Brief Title: Prefrontal Brain Activity and ECG Patterns in Stroke and Healthy Adults
Status: Active, not recruiting | Type: Observational
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Yong-il Shin, Professor, Pusan National University Yangsan Hospital
Other Study IDs: 11-2025-072
Record Dates: First submitted 2025-12-23; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Stroke; Healthy Participants
Keywords: Stroke; Cerebral blood flow; Prefrontal cortex; Electroencephalography (EEG); Functional near-infrared spectroscopy (fNIRS); Electrocardiography (ECG); Healthy Participants
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Intracerebral Hemorrhage (Stroke) Group: Adults with a history of intracerebral hemorrhagic stroke. Participants undergo noninvasive measurements of prefrontal brain activity using fNIRS and EEG, and cardiac activity using ECG, to characterize neurophysiological and electrocardiographic features.
- Cerebral Infarction (Stroke) Group: Adults with a history of cerebral infarction (ischemic stroke). Participants receive the same fNIRS, EEG, and ECG assessments as the hemorrhagic stroke group to compare patterns of brain activation and ECG characteristics.
- Healthy Adult Control Group: Neurologically healthy adults without a history of stroke or major cardiovascular disease. Participants undergo identical fNIRS, EEG, and ECG measurements to serve as a comparison group for stroke patients.

SUMMARY:
This observational study will evaluate brain activity and heart rhythm patterns in people with and without stroke. Brain activity will be measured using functional near-infrared spectroscopy (fNIRS) and electroencephalography (EEG), and cardiac activity will be measured using electrocardiography (ECG). The goal is to characterize differences in prefrontal brain activation and ECG features between stroke patients and healthy adults

DETAILED DESCRIPTION:
This study is an observational investigation designed to characterize neurophysiological and cardiovascular features in adults with a history of stroke and in age-matched healthy controls. Participants will undergo noninvasive measurements of brain activity using functional near-infrared spectroscopy (fNIRS) and electroencephalography (EEG), focusing on prefrontal cortical responses during resting and simple task conditions. Electrocardiography (ECG) will be recorded concurrently to assess heart rate and rhythm characteristics, including temporal and spectral ECG parameters.

The primary objective is to compare patterns of prefrontal brain activation and ECG characteristics between stroke patients and healthy adults, exploring potential associations between altered cortical activity and cardiac autonomic regulation after stroke. Secondary aims include examining relationships between brain signals, ECG features, and clinical factors such as stroke severity or functional status in the patient group. Results from this study may help to generate hypotheses for future interventional research and to identify physiological markers useful for monitoring recovery or risk stratification in stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* Intracerebral Hemorrhage Group (Stroke Patients)

Adults aged 19 to 80 years.

Diagnosed with intracerebral hemorrhage based on clinical evaluation and neuroimaging findings.

Able to read and understand the participant information sheet and consent form, and capable of completing questionnaires in the study language.

Voluntarily agrees to participate in the study, provides written informed consent, and is able to participate for the entire study period.

Cerebral Infarction Group (Stroke Patients)

Adults aged 19 to 80 years.

Diagnosed with cerebral infarction (ischemic stroke) based on clinical evaluation and neuroimaging findings.

Able to read and understand the participant information sheet and consent form, and capable of completing questionnaires in the study language.

Voluntarily agrees to participate in the study, provides written informed consent, and is able to participate for the entire study period.

Healthy Adult Group

Adults aged 19 to 80 years.

No history of stroke or transient ischemic attack (TIA).

No major stroke risk factors such as hypertension, diabetes mellitus, or hyperlipidemia.

No chronic diseases, including cardiovascular disease, chronic kidney disease, or chronic pulmonary disease.

No psychiatric disorders, such as depression or schizophrenia.

Not taking medications that may affect cerebral hemodynamics, including antihypertensive agents, anticoagulants, antiplatelet agents, or antidepressants.

Able to read and understand the participant information sheet and consent form, and capable of completing questionnaires in the study language.

Voluntarily agrees to participate in the study, provides written informed consent, and is able to participate for the entire study period.

Exclusion Criteria:

* Participants meeting any of the following exclusion criteria will not be enrolled in the study.

History of head trauma or cranial surgery within the past 6 months with wounds that have not yet fully healed.

Current diagnosis of a severe psychiatric disorder, such as schizophrenia, major depressive disorder, or bipolar disorder.

Participation in another clinical study and intake of an investigational drug within the past 30 days.

Women who are pregnant or breastfeeding.

Presence of an acute infection or inflammatory disease.

Inability to adequately understand the study procedures or lack of voluntary consent to participate.

Any other clinically significant finding that, in the judgment of the principal investigator or designated study physician, makes the individual unsuitable for participation in this study.

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults aged 19 to 80 years, including patients with intracerebral hemorrhage, patients with cerebral infarction, and neurologically healthy adult volunteers who meet the study's inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Resting-State Prefrontal EEG Activity | Single assessment at one visit (approximately 30-minute session).
  Quantitative characteristics of resting-state electroencephalographic (EEG) activity recorded from the prefrontal cortex (Fp1, Fp2, F7, F8) using a 10-20 electrode placement system during 10 minutes of eyes-closed rest. EEG is obtained once for each participant in one of three groups (intracerebral hemorrhage, cerebral infarction, healthy adults) within a 30-minute session including approximately 10 minutes of preparation, 10 minutes of recording, and 10 minutes of completion procedures.
Resting-State Prefrontal fNIRS Oxygenation | Single assessment at one visit (approximately 30-minute session).
  Changes in oxy-hemoglobin and deoxy-hemoglobin concentrations in the prefrontal cortex (corresponding to Fp1, Fp2, F7, F8) measured by functional near-infrared spectroscopy (fNIRS) during 10 minutes of eyes-closed rest. fNIRS is performed once for each participant in the same 30-minute session (about 10 minutes preparation, 10 minutes recording, 10 minutes completion) in one of the three groups.
Resting-State Electrocardiographic Parameters | Single assessment at one visit (approximately 30-minute session).
  Electrocardiographic (ECG) characteristics recorded for 10 minutes during eyes-closed rest, using electrodes attached to the ears and both wrists, including heart rate, rhythm, and time- and frequency-domain indices of heart rate variability. ECG is measured once for each participant during the same 30-minute session (around 10 minutes preparation, 10 minutes recording, 10 minutes completion) in one of the three groups.

CONTACTS AND LOCATIONS:
Locations (1):
- Rehab lab, Pusan National University Yangsan Hospital, Yangsan, Gyeongsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) cannot be shared due to protection of participants' personal infand regulatory restrictions of our hospital.